CLINICAL TRIAL: NCT03851328
Title: Best Possible Medication History at Universitätsspital Basel (USB)
Brief Title: Best Possible Medication History at USB
Acronym: bpmh@USB
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-00575; qu17Gut
Record Dates: First submitted 2019-02-12; First posted 2019-02-22 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Best Possible Medication History
Keywords: Adverse Drug Events (ADEs); Medication Accuracy; Medication Discrepancy
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: BPMH structured interview — creating a standardized medication list by interviewing patient and/ or relatives according to Best Possible Medication History (BPMH) after patient transfer to medical ward

SUMMARY:
This pilot project investigates the use of a structured medication history (Best Possible Medication History, BPMH) in patients (primarily admitted at the emergency department of University Hospital Basel) after transfer to a medical ward. Unintentional medication discrepancies are analyzed comparing outpatient and inpatient medication therapy.

ELIGIBILITY:
Inclusion Criteria:

* Admission to Emergency Department of University Hospital Basel and transfer to medical ward

Exclusion Criteria:

* medication history taken at Emergency Department of University Hospital Basel not present

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Emergency Department of University Hospital Basel and being transfered to medical ward
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
unintended medication discrepancy | single time point (1 day after admission to hospital)
  number of unintended medication discrepancies comparing medication history taken when admitted to emergency department and BPMH after transfer to medical ward

SECONDARY OUTCOMES:
Categorisation ( Class1, Class2, Class3) for clinical relevance of unintended medication discrepancy | during 7 days after admission to hospital
  expert panel classifies each unintended medication discrepancy in 1 of 3 classes for its potential to cause patient harm. Class 1 discrepancies are those unlikely to cause patient discomfort or clinical deterioration. Class 2 discrepancies could potentially result in moderate discomfort or clinical deterioration. Class 3 discrepancies could potentially result in severe discomfort or clinical deterioration.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Gut, Principal Investigator — Spitalpharmazie Universitätsspital Basel (USB)
Locations (1):
- Spitalpharmazie Universitätsspital Basel (USB), Basel, Switzerland